CLINICAL TRIAL: NCT04201353
Title: Optimizing the Efficiency and Implementation of Cash Transfers to Improve Adherence to Antiretroviral Therapy, Phase II: Effectiveness Study
Brief Title: Optimizing the Efficiency and Implementation of Cash Transfers to Improve Adherence to Antiretroviral Therapy Phase II
Acronym: Afya 2 Phase2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Collaborators: Health for a Prosperous Nation (Other); Rasello (Industry); Tanzania Ministry of Health, Community Development, Gender, Elderly and Children (Unknown)
Responsible Party: Principal Investigator, Sandra McCoy, Associate Professor in Residence, University of California, Berkeley
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: R01MH112432-01A2 (NIH)
Record Dates: First submitted 2019-12-11; First posted 2019-12-17 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: HIV (Human Immunodeficiency Virus)
Keywords: Antiretroviral Treatment Adherence; Conditional Cash Transfers; Tanzania; People Living With HIV; Behavioral Economics
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: 2-arm cluster randomized control trial, with HIV primary care clinic as the unit of randomization
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Facility staff will not be blinded to intervention assignment. However, all other research staff will be blinded to intervention assignment. In addition, participants will not be told during the consent process that as part of the study there are intervention and control clinics. The rationale for this is to prevent patients transferring from intervention to control clinics if they find out that there are some clinics offering cash transfers to new ART clients. Large numbers of transferring patients will compromise the integrity of the study and will create an undue burden for facility staff at intervention clinics.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conditional Cash Transfer (Experimental): Participants attending intervention clinics will have the opportunity to receive up to 6 consecutive monthly cash transfers of 22,500 TSH (~$10) each, conditional on visit attendance with the HIV care provider. Cash transfers will be given once monthly for up to 6 months, spaced ≥25 days apart (consistent with National Guidelines for monthly or bimonthly visits) and are conditional on visit attendance. This means that the cash transfer is only given when the patient visits the clinic for their routine appointment, regardless of whether the visit is earlier or later than the scheduled appointment.
  Interventions: Behavioral: Conditional Cash Transfer
- Control (No Intervention): Participants attending control clinics will receive the standard of care.

INTERVENTIONS:
Behavioral: Conditional Cash Transfer — The intervention is a monthly cash transfer of 22,500 Tanzanian Shillings (~$10) for up to 6 months conditional on visit attendance.
  Arms: Conditional Cash Transfer

SUMMARY:
This protocol describes a 2-arm cluster, randomized controlled trial designed to test the effectiveness of a conditional cash transfer on viral suppression at 12 months post-ART initiation among PHWHIV who have initiated ART within the past 30 days. Randomization will take place at the clinic level (HIV primary care clinics), and eligible participants attending intervention clinics will have the opportunity to receive up to 6 consecutive monthly cash transfers of 22,500 TSH (~$10) each, conditional on visit attendance with the HIV care provider. The study will take place at 32 clinics across four regions in Tanzania: Gaeta, Mwanza, Kagera and Shinyanga. The primary endpoint is viral suppression at 12 months, defined as the proportion of people living with HIV (PLHIV) retained in HIV primary care and with suppressed HIV viral load 12 months after starting ART.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 18 years of age
* Living with HIV infection
* Initiated on antiretroviral therapy less than or equal to 1 month prior to enrollment in the study
* Have access to a mobile phone (ownership, shared ownership, or access to a trusted person's phone)
* Do not intend to transfer to a different facility for HIV care within the following 12 months.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1984 (Actual)
Dates: Start 2020-03-09 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
12-month Viral Suppression | 12 months
  the proportion of people living with HIV (PLHIV) retained in HIV primary care and with suppressed HIV viral load 12 months after starting ART. The primary outcome is expressed as a binary variable, defined as PLHIV who are on ART and with sufficient HIV viral suppression (<1000 copies/ml, WHO's threshold for virologic failure in LMICs) versus not on ART or viral failure (≥1000 copies/ml).

SECONDARY OUTCOMES:
Appointment Attendance | 12 months
  The proportion of scheduled visits that were completed during the 0-12 month period
6-month Viral Suppression | 6 month
  the proportion of people living with HIV (PLHIV) retained in HIV primary care and with suppressed HIV viral load 12 months after starting ART. The primary outcome is expressed as a binary variable, defined as PLHIV who are on ART and with sufficient HIV viral suppression (<1000 copies/ml, WHO's threshold for virologic failure in LMICs) versus not on ART or viral failure (≥1000 copies/ml).
Proportion Virally Suppressed | 12 months
  • The proportion virally suppressed (<1000 copies/ml) of those PLHIV with a viral load result

CONTACTS AND LOCATIONS:
Overall Officials: Sandra McCoy, PhD, Principal Investigator — University of California, Berkeley
Locations (1):
- Health for a Prosperous Nation (HPON), Dar es Salaam, Tanzania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Katabaro E, Joseph B, Mwenda N, Bhattarai P, Msasa J, Mnyippembe A, Maila H, Hassan K, Kunesh J, Sabasaba A, Winters S, Njau P, Hemono R, McCoy SI, Packel L. Scaling-up an mHealth system to deliver financial incentives to improve adherence to antiretroviral therapy in Tanzania. Implement Sci Commun. 2025 Oct 3;6(1):100. doi: 10.1186/s43058-025-00766-1. PMID 41044777
- [Derived] Njau PF, Katabaro E, Winters S, Sabasaba A, Hassan K, Joseph B, Maila H, Msasa J, Fahey CA, Packel L, Dow WH, Jewell NP, Ulenga N, Mwenda N, McCoy SI. Impact of financial incentives on viral suppression among adults initiating HIV treatment in Tanzania: a hybrid effectiveness-implementation trial. Lancet HIV. 2024 Sep;11(9):e586-e597. doi: 10.1016/S2352-3018(24)00149-8. Epub 2024 Aug 1. PMID 39098325
- [Derived] Winters S, Sabasaba A, Fahey CA, Packel L, Katabaro E, Ndungile Y, Njau PF, McCoy SI. Increased prevalence of depression and anxiety among adults initiating antiretroviral therapy during the COVID-19 pandemic in Shinyanga region, Tanzania. AIDS Res Ther. 2023 Jun 10;20(1):36. doi: 10.1186/s12981-023-00534-y. PMID 37301833
- [Derived] Packel L, Njau P, Fahey C, Ramadhani A, Dow WH, Jewell NP, McCoy S. Optimizing the efficiency and implementation of cash transfers to improve adherence to antiretroviral therapy: study protocol for a cluster randomized controlled trial. Trials. 2020 Nov 23;21(1):963. doi: 10.1186/s13063-020-04899-7. PMID 33228757